CLINICAL TRIAL: NCT06162455
Title: High-dose Inhaled NO Therapy for the Prevention of Nosocomial Pneumonia After Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: High-dose Inhaled NO Therapy for the Prevention of Nosocomial Pneumonia After Cardiac Surgery With CPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RECORD Pilot
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Nosocomial Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Oxygen-air mixture without NO after extubation within 5 days after surgery 2 times a day for 30 min
  Interventions: Drug: Sham treatment
- 200 ppm (Experimental): NO will be supplemented at 200-ppm concentration after extubation within 5 days after surgery 2 times a day for 30 min
  Interventions: Drug: 200- ppm NO

INTERVENTIONS:
Drug: Sham treatment — Oxygen-air mixture without NO after extubation after surgery for 5 days 2 times a day for 30 min
  Other Names: Oxygen-Air Mixture
  Arms: Control group
Drug: 200- ppm NO — NO will be supplemented at 200-ppm concentration after surgery for 5 days 2 times a day for 30 min
  Other Names: Nitric Oxide
  Arms: 200 ppm

SUMMARY:
The primary aim of this single-center, prospective, randomized, controlled, pilot study is to test the hypothesis that inhalation of NO 200 ppm prevents the development of nosocomial pneumonia in patients at risk after cardiac surgery with CPB. The study is interventional. Examination and treatment of patients is carried out in accordance with the approved standards of medical care for the relevant diseases. During the study, no experimental or unregistered (not approved for use) medical or diagnostic procedures in the territory of the Russian Federation will be carried out. The study includes patients admitted to the Cardiac Surgery Department of Cardiology Research Institute of Tomsk National Research Medical Center for elective surgery with CPB.

DETAILED DESCRIPTION:
NOSOCOMIAL PNEUMONIA AFTER CARDIAC SURGERY WITH CADIOPULMONARY BYPASS. Nosocomial pneumonia (NP) is one of the most common complications of cardiac surgery with cardiopulmonary bypass (CPB), its frequency according to various sources ranges from 2 to 10% . This complication is accompanied by higher mortality (0.7-4% in patients without pneumonia vs. 25.1-28.2% in patients with pneumonia) , prolonged hospital stay and increased economic costs.

In the retrospective analysis of medical histories of patients operated on CPB for 2020, 2021 and 2022, 3 main risk factors for the development of NP in the postoperative period were identified: time of CPB ≥ 96 minutes, duration of mechanical ventilation ≥ 14 hours, and the presence of atrial fibrillation (AF) before surgery.

STUDY NATURE In relation to medical procedures, this study is observational. The examination and treatment of patients will be carried out in accordance with the approved standards of medical care for the respective diseases. In this study, no experimental or unregistered (not approved for use) medical or diagnostic procedures on the territory of the Russian Federation will be carried out.

STUDY TYPE Single-center, prospective, double-blind, randomized, controlled, parallel group study.

STUDY OBJECTIVES

PRIMARY OBJECTIVE To test the hypothesis that inhalation of NO 200 ppm prevents the development of NP in patients at risk after cardiac surgery with CPB.

SECONDARY OBJECTIVES

1. To test the hypothesis that inhalation of NO 200 ppm twice a day for 30 minutes for 5 days is safe for patients.
2. To compare the level of acute-phase reactants and their dynamics in the main and control groups

RATIONALE FOR RANDOMIZATION There is currently no convincing evidence of benefits or harms of NO inhalation as part of the prevention of NP after cardiac surgery with CPB. Thus, there is no reason to believe that randomization to study groups creates additional risks / benefits for patients. Nevertheless, regardless of the results of randomization, the decision on the possibility of prophylactic NO inhalation after cardiac surgery in each case will be made by a special medical commission consisting of a cardiac surgeon, anesthesiologist and cardiologist, immediately after the patient is enrolled in the study.

PATIENT RANDOMIZATION Patients eligible for this study will be randomized to the intervention group (NO group) and Control group in a 1: 1 ratio according to the randomization sequence generated by a computer program with random numbers by 37 people in each group.

Patients will be randomized immediately after screening and signing the informed consent. Patients in both groups will not receive NO outside of the study protocol until discharged from the hospital. Patient randomization will be performed by a non-blinded NO delivery investigator who is not involved in the clinical management of the patient and the evaluation of treatment outcomes. Patients in the intervention group will receive inhaled NO therapy at a dose of 200 ppm 2 times a day for 5 days or until pneumonia is detected. In the control group, instead of inhaled NO therapy, patients will receive "Sham treatment": similar equipment and observation protocol during the intervention will be used as in the main group, but NO will not be added to the delivered gas mixture.

BLINDING The gas supply systems will look the same for patients of both NO group and Control group. Patients, treating physicians, investigators and other professionals involved in the interpretation of the results will not be aware of the nature of the therapy until the end of the study. The investigating doctor who is responsible for the delivery and monitoring of the investigated gas will remain unblinded and will be responsible for blinding the gas delivery systems, monitoring and securing the delivery, and maintaining the randomization codes. Randomization codes will be sealed in sequentially numbered opaque envelopes. The sequential envelope numbers will serve as randomization numbers that will be recorded in patient's case report form (CRF) and used when necessary, for example, to treat complications.

DOSAGE REGIMEN AND DURATION OF THERAPY

When choosing the dose and timing of NO exposure, clinicians should be guided by 2 basic principles:

1. The dose of NO used and its exposure time must be safe for patients;
2. The dose of NO used and its exposure time must be sufficient to provide potential preventive effects.

NO dosing guidelines for the prevention of pneumonia after cardiac surgery with CPB have not currently been developed, however, there is extensive data from experimental and clinical studies indicating the potential efficacy of a gas concentration of 200 ppm and an exposure time of 30 minutes, which will be implemented in the study.

The safety of using NO for humans in doses of 160-200 ppm for 15-30 minutes 2 to 5 times a day has been demonstrated in a number of clinical studies, including in pregnant women and newborns. The absence of toxic effects of NO at a dose of 200 ppm has been proven on cultured skin fibroblasts, monocytes, macrophages and pulmonary epithelium. Most researchers emphasize the efficacy of intermittent multiple high-dose (160-200 ppm) NO therapy with an average duration of each inhalation for 30 minutes.

NO DELIVERY After screening and signing the informed consent, patients will be randomized into one of the study groups: a control group with sham-treatment and a study group, in which participants will receive inhalation of NO 200 ppm for 30 minutes twice a day for 5 days after extubation and transfer from the intensive care unit. NO delivery will be carried out using a semi-open circuit.

The source of NO is the certified device, which synthesizes NO from atmospheric air using the method of plasma-chemical synthesis directly during therapy. The supply line for the studied gas is built into the supply line for the carrier gas (atmospheric air), the flow of which is provided by a compressor with a maximum flow of 18 l/min, which can be adjusted. The carrier gas flow and NO synthesis rate will be adjusted automatically so that the NO concentration is up to 200 ppm. Next, the gas mixture enters a 3-liter reservoir bag, from where the patient actively breathes it in. To separate the inspiratory and expiratory parts, inhalation and exhalation valves are provided in the circuit. To create an air tight seal with the circuit and patient's airways, correct sized air cushion anesthesia masks will be used. Gas is continuously sampled from the proximal end of the inspiratory part of the circuit to determine the concentration of NO and NO2 in it.

MetHb levels during NO inhalation will be estimated continuously using a peripheral pulse oximeter with fractional saturation capability. During NO therapy, MetHb levels will be maintained at <5%.

NO undergoes a chemical reaction to form NO2, which is an extremely toxic gas and can cause airway inflammation and lung tissue injury. This study regulates the control and maintenance of inhaled NO2 levels below 3 ppm.

During NO therapy, vital functions and safety will be assessed immediately before the initiation of the session, after 15 minutes of NO and after its completion (Heart Rate, Blood Pressure, Respiratory Rate, Oxygen Saturation, MetHb).

In addition, as part of the exploratory endpoint study, exhaled NO levels will be measured immediately before and after inhalation, 10 and 20 minutes after the end of inhalation.

Patients from the control group will undergo sham-treatment, the algorithm of which is similar to inhalation in the main group, but NO will not be added to the gas mixture.

SUMMARY OF KNOWN AND POTENTIAL RISKS AND BENEFITS OF NO-THERAPY NO undergoes a chemical reaction to form NO2. NO2 is an extremely toxic gas that can cause airway inflammation and lung tissue injury. Protocols in use today require that inhaled NO2 levels should be maintained below 3 ppm during NO therapy. The rate of NO2 formation depends on the concentration of NO and O2 in the inhaled gas-air mixture. This fact is important: sources with high concentrations of NO should be avoided; NO and inspiratory fraction of O2 (FiO2) should be used in the minimum clinically acceptable doses. During bench tests of the delivery system, NO2 concentration did not exceed 3 ppm when 200 ppm NO was supplied against the background of FiO2 = 100% (due to the use of a chemical sorbent), however, the minimum sufficient inspiratory fraction of O2 will be used when carrying out the study. NO oxidizes hemoglobin (Hb) (Fe+2) to form (MetHb) (Fe+3), which is unable to transport and release oxygen into the tissue and, as a result, can cause tissue hypoxia. Cyanosis is observed when MetHb levels approach 15-20%. The Institutional Review Board for this study recommended monitoring and maintaining MetHb levels below 5% of total hemoglobin concentration. MetHb levels will be continuously monitored using a peripheral pulse oximeter with the ability to measure fractional saturation (non-invasive pulse co-oximetry). If MetHb levels exceed 5% of the total Hb concentration, NO delivery will be stopped. An increase in MetHb levels > 30% as a critical incident in the study requires intravenous administration of methylene blue in 0.1-0.2 ml/kg of 1% solution (1-2 mg/kg).

After half of the patients are recruited and preliminary statistical analysis is completed, a report on possible complications associated with the potentially negative effects of NO will be submitted.

ASSESSMENT OF CLINICAL EFFECTIVENESS Assessment of clinical effectiveness will be based on the incidence of NP in participants in the study groups.

LABORATORY ASSESSMENT Laboratory efficiency will be assessed by the dynamics of leukocyte and CRP levels.

ASSESSMENT OF INSTRUMENTAL EFFICIENCY Instrumental efficiency will be assessed based on the dynamics of the S/F index and temperature curve.

OBSERVATION PERIOD Monitoring of patients and registration of study data will be carried out until discharge from the hospital. The expected length of hospital stay after uncomplicated cardiac surgery will be approximately 2 weeks.

If complications occur during the perioperative period, patients will be monitored until the event resolves/stabilizes.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac surgery with CPB at current hospitalization.
2. Age > 18 years.
3. Signed informed consent.
4. The presence of at least one risk factor for the development of postoperative NP (CPB time ≥ 96 minutes and/or mechanical ventilation ≥ 14 hours and/or atrial fibrillation before surgery).

Exclusion Criteria:

1. Emergency surgery.
2. Acute coronary syndrome 30 days before surgery.
3. Surgery for active infective endocarditis requiring antibiotic therapy.
4. Diagnosed infectious process of another localization (surgical site infection (SSI), acute and chronic urinary tract infection (active), catheter-related bloodstream infection, peritonitis, etc.).
5. Taking antibacterial drugs for 14 days preceding surgery.
6. Other complications of the postoperative period (pneumothorax requiring pleural drainage, perioperative myocardial infarction accompanied by pulmonary edema, shock of any etiology during the current hospitalization).
7. Potentially dialysis-dependent stage 2 and higher acute kidney injury (according to KDIGO) in the early postoperative period (the criteria for potentially dialysis-dependent acute kidney injury will include patients with stage 2 acute kidney injury and: oliguria against the background of normo-hypervolemia and resistance to loop diuretics and/or oliguria against the background of conducting infusion therapy due to hypovolemia and resistance to loop diuretics).
8. Continued mechanical ventilation.
9. Delirium.
10. Presence of tracheostomy.
11. Patient's participation in another clinical trial at the time of screening or within the previous 3 months.
12. Concomitant pulmonary disease with the need for respiratory support before surgery.
13. History of malignancy or other irreversible diseases/conditions with a 6-month mortality rate >50%.
14. Presence of HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Incidence of nosocomial pneumonia (percent) | From the date of randomization until the date of discharge from hospital (from 2 to 4 weeks)
  Differences between groups in the incidence of nosocomial pneumonia development (percent).

SECONDARY OUTCOMES:
Level of fever (˚C) | 7 days
  The difference in the levels of fever (˚C) between the study groups after the end of the course of inhalations.
Level of leukocytes (counts) | 7 days
  The difference in the levels of leukocytes (10*9/L) between the study groups after the end of the course of inhalations.
Level of C-reactive protein (mg/L) | 7 days
  The difference in the levels of C-reactive protein (CRP) (mg/L) between the study groups after the end of the course of inhalations.
S/F index (ratio) | 7 days
  Change in the ratio of oxygen saturation to inspiratory oxygen fraction (S/F index) in the study groups between day 7 and the day of randomization.
Incidence of sepsis and septic shock (percent) | 7 days
  Difference in the incidence of sepsis and septic shock during hospitalization in patients of both groups (percent).
Incidence of extrapulmonary complications (percent) | 7 days
  Difference in the incidence of extrapulmonary complications between the study groups (percent).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay O. Kamenshchikov, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute Tomsk National Research Medical Center, Tomsk, Select..., Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF)
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.